CLINICAL TRIAL: NCT00241618
Title: Phase IV Study of Treatment of Acute Hepatitis C With Pegylated Interferon
Brief Title: Timing and Duration of Acute Hepatitis C Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: University Hospital Freiburg (Other); Beth Israel Deaconess Medical Center (Other); Alexander von Humboldt Association (Other); Fulbright (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Tempus AI (Industry); International Society for Infectious Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 994058402; AI054887; AI41563; Fulbright; TEMPUS; ISID
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Hepatitis C
Keywords: Clinical trial; Randomized; Treatment; Prospective; Parallel Assignment; Efficacy Safety Study
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alpha 2
Drug: Ribavirin

SUMMARY:
Spontaneous resolution of acute hepatitis C infection cannot be predicted and the majority of cases persist and become chronic. This randomized trial assesses the efficacy and safety of peginterferon alfa-2b. The investigators hypothesize that therapy strategies could prevent the development of chronic hepatitis.

DETAILED DESCRIPTION:
With nearly 4 million people in the United States, and an estimated 170-200 million people worldwide, the hepatitis C virus (HCV) represents a clear and significant public health issue. Unfortunately, for most people infected with HCV (70%-85%) spontaneous resolution is uncommon and 60% to 80% of patients with acute hepatitis C infection develop chronic hepatitis. This randomized trial focuses on defining the effect of treatment of acute HCV on prevention of chronic hepatitis in addition to optimization of the treatment regimen, onset and the length of peginterferon alpha therapy in acute hepatitis C infections. This randomized, multi-center prospective study assesses the efficacy of peginterferon in acute hepatitis. We will also compare differences in sustained viral response rates in patients with acute hepatitis C starting treatment at 8, 12, or 24 weeks. We will also compare the efficacy of 8, 12 or 24 weeks therapy with PEG-IFN-alpha. All eligible patients are enrolled and screened for an initial observation period starting from the time of their first positive HCV-RNA-PCR, during which bi-weekly serum ALT and HCV-RNA subjects were performed. Patients who did not resolve spontaneously (loss of HCV-RNA without treatment) by the end of the observation period were randomly assigned to receive PEG-IFN-alpha at the assigned onset and/or duration. Patients who do not consent to therapy at enrollment are included as a non-randomized comparison group. All subjects with SVR were followed for 48 weeks after the follow-up at 24 weeks when SVR was determined.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-50 years, with or without symptoms
* Diagnosis of acute hepatitis C: elevated serum alanine aminotransferase (ALT) > 10 times the upper limit of normal (ULN)
* Seroconversion from negative to positive anti-HCV antibody status (third-generation enzyme-linked immunosorbent assay)
* Conversion from negative to positive polymerase chain reaction (PCR) for HCV-RNA, ruling out other causes of hepatitis by history and appropriate serologic and virologic studies.

Exclusion Criteria:

* Decompensated liver disease
* Coinfection with human immunodeficiency virus (HIV) or Schistosoma mansoni
* Marked anemia (hemoglobin level ≤ 120 g/L in women and ≤ 130 g/L in men)
* Neutropenia (< 1,500/mm3)
* Thrombocytopenia (< 90,000/mm3)
* A creatinine concentration > 1.5 times ULN
* Serum alpha-fetoprotein > 25 ng/ml
* An organ transplant
* Neoplastic disease
* Severe cardiac or pulmonary disease
* Unstable thyroid dysfunction
* A psychiatric disorder
* Seizure disorder
* Severe retinopathy
* A current pregnancy or were breast feeding or unwillingness to practice contraception
* Therapy with immunomodulatory agents within the last 6 months
* Alcohol or drug dependence within 1 year of study entry.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180
Dates: Start 2002-01; Study Completion 2006-01

PRIMARY OUTCOMES:
Sustained viral response rate in treatment group versus control

SECONDARY OUTCOMES:
End of treatment virologic response
Early virologic response at week 4
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Ismail, M.D., Study Chair — Ain Shams University; Sanaa M Kamal, M.D., Principal Investigator — Ain Shams University; Nezam H Afdhal, M.D., Principal Investigator — Harvard Medical School (HMS and HSDM); Manal El Sayed, M.D., Principal Investigator — ASU
Locations (3):
- Egypt (3):
  - ASU Specialized Hospital, Cairo, Cairo Governorate
  - ASU, Cairo
  - Shebin Liver Center, Cairo

REFERENCES:
- [Background] Kamal SM, Ismail A, Graham CS, He Q, Rasenack JW, Peters T, Tawil AA, Fehr JJ, Khalifa Kel S, Madwar MM, Koziel MJ. Pegylated interferon alpha therapy in acute hepatitis C: relation to hepatitis C virus-specific T cell response kinetics. Hepatology. 2004 Jun;39(6):1721-31. doi: 10.1002/hep.20266. PMID 15185314
- [Background] Gerlach JT, Diepolder HM, Zachoval R, Gruener NH, Jung MC, Ulsenheimer A, Schraut WW, Schirren CA, Waechtler M, Backmund M, Pape GR. Acute hepatitis C: high rate of both spontaneous and treatment-induced viral clearance. Gastroenterology. 2003 Jul;125(1):80-8. doi: 10.1016/s0016-5085(03)00668-1. PMID 12851873
- [Background] Nomura H, Sou S, Tanimoto H, Nagahama T, Kimura Y, Hayashi J, Ishibashi H, Kashiwagi S. Short-term interferon-alfa therapy for acute hepatitis C: a randomized controlled trial. Hepatology. 2004 May;39(5):1213-9. doi: 10.1002/hep.20196. PMID 15122749
- [Background] Kamal SM, Rasenack JW, Bianchi L, Al Tawil A, El Sayed Khalifa K, Peter T, Mansour H, Ezzat W, Koziel M. Acute hepatitis C without and with schistosomiasis: correlation with hepatitis C-specific CD4(+) T-cell and cytokine response. Gastroenterology. 2001 Sep;121(3):646-56. doi: 10.1053/gast.2001.27024. PMID 11522749
- [Background] Santantonio T, Sinisi E, Guastadisegni A, Casalino C, Mazzola M, Gentile A, Leandro G, Pastore G. Natural course of acute hepatitis C: a long-term prospective study. Dig Liver Dis. 2003 Feb;35(2):104-13. doi: 10.1016/s1590-8658(03)00007-0. PMID 12747629
- [Background] Wiegand J, Jackel E, Cornberg M, Hinrichsen H, Dietrich M, Kroeger J, Fritsch WP, Kubitschke A, Aslan N, Tillmann HL, Manns MP, Wedemeyer H. Long-term follow-up after successful interferon therapy of acute hepatitis C. Hepatology. 2004 Jul;40(1):98-107. doi: 10.1002/hep.20291. PMID 15239091
- [Background] Kamal SM, El Tawil AA, Nakano T, He Q, Rasenack J, Hakam SA, Saleh WA, Ismail A, Aziz AA, Madwar MA. Peginterferon alpha-2b and ribavirin therapy in chronic hepatitis C genotype 4: impact of treatment duration and viral kinetics on sustained virological response. Gut. 2005 Jun;54(6):858-66. doi: 10.1136/gut.2004.057182. PMID 15888797
- [Background] Jaeckel E, Cornberg M, Wedemeyer H, Santantonio T, Mayer J, Zankel M, Pastore G, Dietrich M, Trautwein C, Manns MP; German Acute Hepatitis C Therapy Group. Treatment of acute hepatitis C with interferon alfa-2b. N Engl J Med. 2001 Nov 15;345(20):1452-7. doi: 10.1056/NEJMoa011232. PMID 11794193
- [Background] Larghi A, Zuin M, Crosignani A, Ribero ML, Pipia C, Battezzati PM, Binelli G, Donato F, Zanetti AR, Podda M, Tagger A. Outcome of an outbreak of acute hepatitis C among healthy volunteers participating in pharmacokinetics studies. Hepatology. 2002 Oct;36(4 Pt 1):993-1000. doi: 10.1053/jhep.2002.36129. PMID 12297849